CLINICAL TRIAL: NCT06818084
Title: Transcatheter Treatment of Pure Aortic Regurgitation With VitaFlow Liberty System: a Prospective, Multicenter Study
Brief Title: TRanscAtheter TreatMent of PurE Aortic Regurgitation With VitaFlow Liberty System
Acronym: TRAMPERS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhu zhengbin, Principal Investigator, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24SF1904800; 24SF1904800 (Other: Shanghai Science & Technology Commission)
Record Dates: First submitted 2025-01-25; First posted 2025-02-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: AORTIC VALVE DISEASES; Aortic Regurgitation; Transcatheter Aortic Valve Replacement (TAVR)
Keywords: pure aortic regurgitation; Transcatheter aortic valve replacement (TAVR); hypoattenuated leaflet thickening; reduced leaflet motion
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VitaFlow (Experimental): Patients who meet the inclusion and exclusion criteria will undergo TAVR using the VitaFlow™ self-expanding valve system.
  Interventions: Combination Product: VitaFlow+GDMT
- J-Valve (Active Comparator): Patients who meet the inclusion and exclusion criteria will undergo TF-TAVR using dedicated transcatheter device J-Valve system.
  Interventions: Combination Product: J-Valve+GDMT

INTERVENTIONS:
Combination Product: VitaFlow+GDMT — The patient will undergo transcatheter aortic valve replacement on the basis of guideline-directed medical therapy with The VitaFlow™ system.
  The VitaFlow™ system (MicroPort®, Shanghai, China) was a novel TAVR system, which incorporates high-radial force and a double layer polyethylene terephthalate (PET) skirt to optimize frame geometry and minimize the risks of paravalvular leak (PVL). The VitaFlow™ transcatheter aortic valve is made of a self-expanding nitinol frame and tri-leaflet bovine pericardial valve.
  Arms: VitaFlow
Combination Product: J-Valve+GDMT — The patient will undergo transfemoral aortic valve replacement on the basis of guideline-directed medical therapy with The J-Valve system (Jie ChengMedical Technologies, Suzhou, China). The J-Valve system is a second-generation self-expand able device composed of a porcine bioprosthetic aortic valve and a transfemoral delivery sheath. The valve is supported by a self-expanding nitinol structure. The different valve sizes are 21, 23, 25, 27, 29 and 34 mm. Three U-shaped nitinol graspers were designed to surround the valve.
  Arms: J-Valve

SUMMARY:
This study is a prospective, multicenter, non-randomized controlled trial, planning to enroll 180 patients with pure native aortic regurgitation. On the basis of standardized medical therapy, patients will be assigned in a 1:1 ratio to undergo transfemoral transcatheter aortic valve replacement (TF-TAVR) . This prospective, multicenter trial aims to evaluate the safety and effectiveness of transfemoral TAVR using the VitaFlow™ self-expanding valve system compared to dedicated transcatheter devices in patients with PNAR.

The primary endpoint is a composite of all-cause mortality, disabling stroke, and rehospitalization for heart failure, myocardial Infarction, and requiring dialysis or valve reoperation at 12 months post-procedure.

Secondary endpoints include procedure-related complications, long-term clinical events, patient functional status and quality of life, bioprosthetic valve imaging follow-up, echocardiographic parameters, and treatment costs. All endpoint definitions conform to the Valve Academic Research Consortium-3 (VARC-3) criteria

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of TF-TAVR for the treatment of isolated aortic regurgitation. The study will compare all-cause mortality, cardiovascular mortality, stroke, rehospitalization for heart failure, and renal failure requiring dialysis treatment at 12 months after TAVR. Additionally, the study will assess the incidence of hypoattenuated leaflet thickening (HALT) and reduced leaflet motion (RLM) via CTA, as well as the aortic valve root-prosthesis coaxiality. Changes and differences between groups in the following parameters will be evaluated using transthoracic echocardiography at 6 and 12 months after enrollment: left ventricular ejection fraction (Simpson method), left ventricular end-diastolic volume index (LVEDVi), left ventricular end-systolic volume index (LVESVi), left ventricular end-diastolic diameter (LVEDd), left ventricular end-systolic diameter (LVESd), estimated aortic valve orifice area, valvular regurgitation, and transvalvular pressure gradient compared with baseline. The study will also compare changes and differences between groups in the Minnesota Living with Heart Failure Questionnaire, Social Support Rating Scale (SSRS), International Physical Activity Questionnaire (IPAQ), and 6-minute walk test (6MWT) at 6 and 12 months after enrollment compared with baseline. Furthermore, the study will compare surgical costs, potential complication costs, and disease-related costs between the two groups.

ELIGIBILITY:
Inclusion Criteria Age ≥ 60 years. Symptomatic moderate-to-severe or greater isolated aortic regurgitation.

Asymptomatic moderate-to-severe or greater isolated aortic regurgitation meeting at least one of the following criteria:

LVEF ≤ 55% (measured by biplane Simpson's method); LVESD > 50 mm ; LVESDi > 22 mm/mm²； LVESVi > 45mL/m2 Anatomical suitability for TAVR as assessed by the heart team. Provision of written informed consent by the patient or their legal guardian, with agreement to the treatment plan and willingness and ability to comply with all required follow-up assessments.

Exclusion Criteria Incomplete coronary revascularization. Less than 30 days of guideline-directed medical therapy at maximally tolerated doses.

Life expectancy < 1 year. LVEF < 45%. eGFR < 30 mL/min/1.73m². Known allergy or contraindication to required medications (e.g., aspirin, clopidogrel, warfarin) or contrast media.

Any condition that precludes contrast-enhanced CT. Concurrent moderate-to-severe or severe valvular heart disease other than aortic regurgitation.

Poor patient compliance, unable to complete follow-up as required. Any other condition that, in the investigator's judgment, would make the patient unsuitable for the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical worsening | 12 months
  The primary endpoint is a composite of all-cause mortality, disabling stroke, and rehospitalization for heart failure, myocardial Infarction, and requiring dialysis or valve reoperation at 12 months post-procedure.

SECONDARY OUTCOMES:
Rate of procedural complications | 12 months
  The rate of any aortic dissection, annular rupture, coronary artery occlusion, vascular complications, permanent pacemaker implantation, reoperation of heart valve.
6-minute walk distance | 12 months
  This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
New York Heart Association (NYHA) functional class | 12 months
  Classification of function capacity of the NYHA.
Rate of hypoattenuated leaflet thickening | 12 months
  The rate of hypoattenuated leaflet thickening. Hypoattenuated leaflet thickening（HALT）defined by VARC-3
Rate of reduced leaflet motion | 12 months
  Rate of reduced leaflet motion. Reduced leaflet motion（RLM）defined by VARC-3.
Rate of Stroke | 12 months
  Stroke is defined as an acute episode of focal or global neurological dysfunction caused by the brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction.
Mortality | 12 months
  All-cause, cardiovascular, and non-cardiovascular mortality
Rate of bleeding complications | 12 months
  Rate of bleeding complications. The original VARC definitions with BARC classifications
Rate of prothetic valve dysfunction | 12 months
  The rate of any prothetic aortic valve stenosis, prothesis-patient mismatch, prosthetic aortic valve regurgitation
Rate of rehospitalization | 12 months
  The rate of rehospitalization due to valve-related symptoms or worsening congestive heart failure.
Quality of life assessment (Minnesota Living with Heart Failure Questionnaire, MLHFQ) | 12 months
  Total score of Minnesota Living with Heart Failure Questionnaire (MLHFQ). The total score ranges from 0 to 105, with higher scores indicating a greater impact of heart failure on quality of life and worse outcome..
Quality of life assessment (social supporting raing scal, SSRS) | 12 months
  Total score of social supporting raing scal (SSRS). The total score ranges from 0 to 40, with higher scores indicating a higher level of social support.
Quality of life assessment (International Physical Activity Questionnaire, IPAQ) | 12 months
  Total score of International Physical Activity Questionnaire (IPAQ). The total score is calculated by multiplying the frequency and duration of each activity by its respective MET value, and then summing these products. The result is a measure of the total energy expenditure from physical activity in MET-minutes per week.The total score can be used to classify individuals into different physical activity levels, such as low, moderate, or high.
Treatment costs | 12 months
  Including surgical costs, potential complications costs, and disease-related costs

OTHER OUTCOMES:
Left ventricular ejection fraction (Simpson's method) | 12 months
  Transthoracic echocardiography measurement of left ventricular ejection fraction (Simpson's method).
  Unit: %
Left ventricular end-diastolic volume index | 12 months
  Transthoracic echocardiography measurement left ventricular end-diastolic volume index (LVEDVi).
  Unit: milliliters per square meter (mL/m²)
Left ventricular end-systolic volume index | 12 months
  Transthoracic echocardiography measurements of left ventricular end-systolic volume index (LVESVi).
  Unit: milliliters per square meter (mL/m²)
Left ventricular end-diastolic diameter | 12 months
  Transthoracic echocardiography measurements of left ventricular end-diastolic diameter (LVEDd).
  Unit: millimeters
Left ventricular end-systolic diameter | 12 months
  Transthoracic echocardiography measurements of left ventricular end-systolic diameter (LVESd).
  Unit: millimeters
Aortic valve orifice area | 12 months
  Transthoracic echocardiography measurement of aortic valve orifice area. Unit: square centimeters
Transvalvular pressure gradient of aortic valve | 12 months
  Transthoracic echocardiography measurement of transvalvular pressure gradient of aortic valve.
  Unit: mmHg

CONTACTS AND LOCATIONS:
Overall Officials: ZhengBin Zhu, MD. PhD, Principal Investigator — Ruijin Hospital
Locations (4):
- China (4):
  - Ruijin hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided